CLINICAL TRIAL: NCT02613429
Title: Identification of Airway Structures Necessary for Airway Access Via the Skin to be Used in Case of Failure to Maintain Oxygenation With Non-invasive Methods
Brief Title: Identification of Airway Structures Necessary for Airway Access Via the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Head of clinical anaesthesia and research, ENT and max fax, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Seventh floor 15/1
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Upper Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranial horizontal (Active Comparator): identification of the airway by from the cranial end. Marking of the airway, including the cricothyroid membrane, on the skin, by starting the examination from the cranial end at the level of the thyroid catilage , horizontally and thereafter moving caudally
  Interventions: Behavioral: identification of the airway by from the cranial end
- caudal longitudinal (Active Comparator): identification of the airway from the distal end. Marking of the airway, including the cricothyroid membrane, on the skin, by starting the examination caudally, and then moving cranially
  Interventions: Behavioral: identification of the airway from the distal end

INTERVENTIONS:
Behavioral: identification of the airway by from the cranial end — The airway is identified with inspection and imaging technique (ultrasound) by placing the ultrasound transducer over the thyroid cartilage and from there moving distally
  Arms: Cranial horizontal
Behavioral: identification of the airway from the distal end — The airway is identified with inspection and imaging technique (ultrasound) by placing the ultrasound transducer over the distal trachea and moving cranially
  Arms: caudal longitudinal

SUMMARY:
Literature shows that anaesthetists have a low success-rate when trying to access the airway percutaneously in case of failed ventilation and intubation.

The study will investigate anaesthetists ability to locate the trachea and the thyroid cartilage and the cricoid cartilage in patients, using different methods including application of ultrasonography.

DETAILED DESCRIPTION:
Literature shows that anaesthetists have a low success-rate when trying to access the airway percutaneously in case of failed ventilation and intubation.

The researchers will investigate anaesthetists ability to locate the trachea and the thyroid cartilage and the cricoid cartilage of a healthy subject with different methods including application of ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesiologist

Exclusion Criteria:

* unvillingnes to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
time to identify the structures necessary for percutaneous airway acess | two minutes after initiation of the attempt to identify the airway structures

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, M.D., Study Chair — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, department of anaesthesia, Copenhagen
  - Rigshospitalet, section for anaesthesia for ENT and Maxillofacial surgery, section 3071, Copenhagen